CLINICAL TRIAL: NCT02004665
Title: Incidence and Prognostic Value of DELIRIUM in Patients With Acute CORonary synDrome: an observatIonal Study by the DELIRIUM-CORDIS Investigators.
Brief Title: Incidence and Prognostic Value of DELIRIUM in Patients With Acute CORonary synDrome: an observatIonal Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale San Donato (Other)
Responsible Party: Principal Investigator, Leonardo Bolognese, MD, Director, Ospedale San Donato
Other Study IDs: Arezzo012
Record Dates: First submitted 2013-11-24; First posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Delirium; Acute Coronary Syndrome
MeSH Terms: conditions — Delirium; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- acute coronary syndrome and delirium: patients with acute coronary syndrome and delirium

SUMMARY:
to evaluate the incidence of delirium in patients with acute coronary syndrome and its correlation with adverse events

ELIGIBILITY:
Inclusion Criteria:

* acute coronary syndrome patients undergone coronary revascularization or referred to conservative strategy
* age ≥ 70 years
* diagnosis of delirium by the Confusion Assessment Method in the ICU (CAM-ICU) scale

Exclusion Criteria:

* none

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients with acute coronary syndrome and delirium
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
in-hospital adverse events incidence | until discharge (4-7 days from admission)

SECONDARY OUTCOMES:
12-month adverse events incidence | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Department, Ospedale S.Donato, Arezzo, AR, Italy

REFERENCES:
- [Derived] Falsini G, Grotti S, Porto I, Toccafondi G, Fraticelli A, Angioli P, Ducci K, Liistro F, Pieroni M, Taddei T, Romanelli S, Rossi R, Bolognese L. Long-term prognostic value of delirium in elderly patients with acute cardiac diseases admitted to two cardiac intensive care units: a prospective study (DELIRIUM CORDIS). Eur Heart J Acute Cardiovasc Care. 2018 Oct;7(7):661-670. doi: 10.1177/2048872617695235. Epub 2017 Mar 16. PMID 29064263